CLINICAL TRIAL: NCT05396690
Title: Safety and Efficacy of Remimazolam in Induction and Maintenance of General Anesthesia in OPCAB Surgery
Brief Title: Safety and Efficacy of Remimazolam in OPCAB Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Jiyoung Yoo, associate professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AJIRB-MED-INT-21-641
Record Dates: First submitted 2022-04-15; First posted 2022-05-31 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Coronary Artery Bypass Surgery
MeSH Terms: interventions — remimazolam; Sevoflurane

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- remimazolam group (Experimental): In the Remimazolam group as an induction dose 6 mg/kg/h of remimazolam with 0.5-1.0 mcg/kg of sufentanil was injected together. If consciousness was lost, rocumerone 1 mg/kg was given intravenously, and endotracheal intubation was performed when sufficient muscle relaxation was achieved 2 minutes later.
  Maintenance of anesthesia is achieved by using a programmed infusion pump with remimazolam 1 mg/kg/h (up to 2 mg/kg/h) and sufentanil effect site concentration of 0.4 to 0.5 to reach the appropriate depth of anesthesia. The optimal level of anesthesia is based on maintaining a bispectral index (BIS) of 35-65.
  Interventions: Drug: Remimazolam Injection [Byfavo]
- sevoflurane group (Other): After injection of 2-5 mg of midazolam and 0.5-1.0 mcg/kg of sufentanil as an induction dose, 1 mg/kg of rocumerone is given intravenously when consciousness is lost, and endotracheal intubation is performed when sufficient muscle relaxation is achieved 2 minutes later. For maintenance of anesthesia, the concentration of sevoflurane and sufentanil effect site concentration is 0.4 to 0.5 to reach the appropriate depth of anesthesia, and the optimal degree of anesthesia is based on maintaining the BIS 35 to 65.
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Remimazolam Injection [Byfavo] — Induction dose: 6 mg/kg/h with sufentanil Maintenance dose: 1~2 mg/kg/h with sufentanil If arousal occurs during surgery, rapidly increase the infusion rate of remimazolam to 12 mg/kg/h and infuse for 1 minute. If the patient's arousal persists after these measures, stop remimazolam infusion and replace with another drug.
  Arms: remimazolam group
Drug: Sevoflurane — Induction dose: 2~3 mg midazolam with sufentanil Maintenance: Adjust the concentration to be BIS 35-65 based on 0.5 mac If arousal occurs during surgery, raise the concentration of sevoflurane to 1.5 MAC (increase the total gas flow rate to 8 l/min) and if arousal persists after 1 minute, administer midazolam 2-3 mg.
  Arms: sevoflurane group

SUMMARY:
Remimazolam is a novel short-acting benzodiazepine drug that acts on the benzodiazepine binding site of gamma-aminobutryic acid (GABA) A receptor, is metabolized by esterase, and has a context-sensitive half-time of about 6-7 minutes. Looking at some previous studies using Remimazolam, the safety and efficacy as a general anesthetic have been sufficiently proven.

In particular, compared to intravenous anesthetic agents such as propofol, the action time of anesthetics is relatively longer, but the frequency of hypotension is low. However, most studies have been conducted on patients of American Society Anesthesiologist (ASA) class I-II, and studies on patients with high severity have not yet been sufficiently secured.

Therefore, this study aims to compare the efficacy and safety of Remimazolam as an anesthetic with Sevoflurane in terms of hemodynamics in patients with high severity undergoing OPCAB surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 19 years of age or older to receive OPCAB surgery
* Clinical diagnosis of coronary artery obstructive disease

Exclusion Criteria:

* Ejection fraction < 35% at preoperative ECHO test
* Mitral regurgitation > grade 2 at preoperative ECHO test
* Currently using inotropics
* Currently receiving mechanical support

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2022-06-15 (Estimated); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
cardiac index (T4) | 5 minutes before operation
  The cardiac index (CI) at that time was measured and compared between the two groups.
cardiac index (T5) | 10 minutes after starting left internal mammary artery dissection
  The cardiac index (CI) at that time was measured and compared between the two groups.
cardiac index (T6) | 10 minutes after starting left anterior descending coronary artery anastomosis
  The cardiac index (CI) at that time was measured and compared between the two groups.
cardiac index (T7) | 10 minutes after starting Y-graft anastomosis of graft vessels
  The cardiac index (CI) at that time was measured and compared between the two groups.

SECONDARY OUTCOMES:
NE dose | During surgery(from induction of anesthesia to end of surgery)
  total amount of norepinephrine during OPCAB
Incidence of hypotension | During surgery(from induction of anesthesia to end of surgery)
  The incidence of hypotension during OPCAB are counted by number which based on the anesthetic record.

CONTACTS AND LOCATIONS:
Locations (1):
- Ajou University Hospital, Suwon, Gyeonggido, South Korea